CLINICAL TRIAL: NCT00887822
Title: A Double-Blind, Randomized, Multicenter, Phase III Study of Bevacizumab in Combination With Capecitabine and Cisplatin Versus Placebo in Combination With Capecitabine and Cisplatin, as First-Line Therapy in Patients With Advanced Gastric Cancer.
Brief Title: A Study of Bevacizumab (Avastin) Versus Placebo in Combination With Capecitabine (Xeloda) and Cisplatin as First-Line Therapy for Advanced Gastric Cancer
Acronym: AVATAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML22367
Record Dates: First submitted 2009-04-22; First posted 2009-04-24 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Bevacizumab; Capecitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Bevacizumab, Capecitabine and Cisplatin (Experimental): Participants will receive bevacizumab 7.5 milligrams per kilogram (mg/kg) intravenous (IV) infusion on Day 1 of every 3-week cycle in combination with capecitabine 1000 milligrams per square meter (mg/m^2) orally twice daily (total daily dose 2000 mg/m^2) on Days 1-14 of every 3-week cycle and cisplatin 80 mg/m^2 IV infusion on Day 1 of every 3-week cycle for a maximum of 6 cycles; until disease progression or unmanageable toxicity.
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Cisplatin
- Placebo, Capecitabine and Cisplatin (Placebo Comparator): Participants will receive placebo matched to bevacizumab on Day 1 of every 3-week cycle in combination with capecitabine 1000 mg/m^2 orally twice daily (total daily dose 2000 mg/m^2) on Days 1-14 of every 3-week cycle and cisplatin 80 mg/m^2 IV infusion on Day 1 of every 3-week cycle for a maximum of 6 cycles; until disease progression or unmanageable toxicity.
  Interventions: Drug: Placebo; Drug: Capecitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Bevacizumab — 7.5 mg/kg IV infusion on Day 1 of every 3-week cycle
  Other Names: Avastin
  Arms: Bevacizumab, Capecitabine and Cisplatin
Drug: Placebo — Placebo matched to bevacizumab on Day 1 of every 3-week cycle
  Arms: Placebo, Capecitabine and Cisplatin
Drug: Capecitabine — 1000 mg/m^2 orally twice daily on Days 1-14 of every 3-week cycle
  Other Names: Xeloda
Drug: Cisplatin — 80 mg/m^2 IV infusion on Day 1 of every 3-week cycle for a maximum of 6 cycles

SUMMARY:
This 2 arm study will compare the efficacy and safety of bevacizumab in combination with capecitabine and cisplatin versus placebo in combination with capecitabine and cisplatin in participants who have not received prior chemotherapy for advanced or metastatic gastric cancer. Participants will be randomized to one of two treatment groups Bevacizumab + Capecitabine/Cisplatin (experimental arm) or Placebo + Capecitabine/Cisplatin (control arm).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach or gastro-oesophageal junction with inoperable, locally advanced or metastatic disease, not amenable to curative therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2
* Measurable disease or non-measurable but evaluable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST)

Exclusion Criteria:

* Previous chemotherapy for locally advanced or metastatic gastric cancer
* Previous platinum or anti-angiogenic therapy
* Radiotherapy within 28 days of randomization
* Evidence of Central Nervous System (CNS) metastasis at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- China (9):
  - Beijing
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Shantou
  - Shenyang
  - Wuhan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study reported data up to clinical cut-off date 13 May 2011, as approximately half of the participants withdrew the study at clinical cut-off date. Ad hoc analysis was done for overall survival, with clinical cut-off date of 12 January 2012, subsequent to clinical cut-off date of 13 May 2011.
Groups:
- Bevacizumab, Capecitabine and Cisplatin: Participants received bevacizumab 7.5 milligrams per kilogram (mg/kg) intravenous (IV) infusion on Day 1 of every 3-week cycle in combination with capecitabine 1000 milligrams per square meter (mg/m^2) orally twice daily (total daily dose 2000 mg/m^2) on Days 1-14 of every 3-week cycle and cisplatin 80 mg/m^2 IV infusion on Day 1 of every 3-week cycle for a maximum of 6 cycles; until disease progression or unmanageable toxicity.
- Placebo, Capecitabine and Cisplatin: Participants received placebo matched to bevacizumab on Day 1 of every 3-week cycle in combination with capecitabine 1000 mg/m^2 orally twice daily (total daily dose 2000 mg/m^2) on Days 1-14 of every 3-week cycle and cisplatin 80 mg/m^2 IV infusion on Day 1 of every 3-week cycle for a maximum of 6 cycles; until disease progression or unmanageable toxicity.
Period: Overall Study
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Started | 100 | 102
Treated (Safety Population) | 100 | 101
Completed | 3 | 0
Not Completed | 97 | 102
Not completed — Insufficient therapeutic response | 53 | 55
Not completed — Adverse Event | 14 | 17
Not completed — Failure to return | 11 | 11
Not completed — Refused treatment/Did not cooperate | 12 | 10
Not completed — Administrative/Other than specified | 5 | 4
Not completed — Death | 2 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Bevacizumab, Capecitabine and Cisplatin: Participants received bevacizumab 7.5 mg/kg IV infusion on Day 1 of every 3-week cycle in combination with capecitabine 1000 mg/m^2 orally twice daily (total daily dose 2000 mg/m^2) on Days 1-14 of every 3-week cycle and cisplatin 80 mg/m^2 IV infusion on Day 1 of every 3-week cycle for a maximum of 6 cycles; until disease progression or unmanageable toxicity.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin | Total
Number analyzed (Participants) | 100 | 102 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.66) | 55.5 (12.14) | 54.9 (11.89)
Gender [Count of Participants; unit: Participants]
  Female | 32 | 28 | 60
  Male | 68 | 74 | 142

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Event (Death)
Description: Percentage of participants who died due to any cause was reported. As planned, ad hoc analysis was done for overall survival up to clinical cut-off date of 12 January 2012 (34 months), subsequent to the protocol-defined clinical cut-off date of 13 May 2011 (26 months). Overall survival was defined as the time between randomization and the date of death due to any cause.
Time Frame: From randomization until death (up to 34 months)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
percentage of participants | 77.0 | 75.5

2. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time between randomization and the date of death due to any cause. Overall survival was estimated using Kaplan Meier method. Reported data included censored observations. Participants for whom no death was captured on the clinical database were censored at the most recent date they were known to be alive. As planned, ad hoc analysis was done for overall survival up to clinical clinical cut-off date of 12 January 2012 (34 months), subsequent to the protocol-defined clinical cut-off date of 13 May 2011 (26 months).
Time Frame: From randomization until death (up to 34 months)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
months | 10.5 [8.9 to 14.1] | 11.4 [8.6 to 14.6]
Statistical Analysis 1: Comparison: Bevacizumab, Capecitabine and Cisplatin vs Placebo, Capecitabine and Cisplatin; Test type: Superiority or Other; p = 0.8636, Log Rank; The difference in distribution of survival between the two treatment arms was tested with a two-sided unstratified log-rank test; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.75 to 1.41] — The hazard ratio between the two treatment arms was estimated with a univariate Cox's proportional hazards model

3. Secondary Outcome: Percentage of Participants With Progression-Free Survival (PFS) Events (Disease Progression/Death)
Description: Progression of disease was defined as at least 20 percent (%) increase in the sum of longest diameters of target lesions compared to the smallest sum of longest diameters on-study and absolute increase of at least 5 millimeters (mm), progression of existing non-target lesions, or presence of new lesions. PFS was defined as the time between randomization and the date of first documented disease progression or death, whichever occurred first, according to Response Evaluation Criteria In Solid Tumors (RECIST).
Time Frame: From randomization until disease progression or death (up to 26 months)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
percentage of participants | 81.0 | 81.4

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time between randomization and the date of first documented disease progression or death, whichever occurred first, according to RECIST. Progression of disease was defined as at least 20% increase in the sum of longest diameters of target lesions compared to the smallest sum of longest diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. PFS was estimated using Kaplan Meier method. Reported data included censored observations. Participants who had neither progressed nor died at the time of study completion or who were lost to follow-up were censored at the date of the last tumor assessment or last follow-up for progression of disease. Participants for whom no post-baseline tumor assessments were available were censored at day of randomization.
Time Frame: From randomization until disease progression or death (up to 26 months)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
months | 6.3 [5.7 to 7.4] | 6.0 [4.9 to 7.4]
Statistical Analysis 1: Comparison: Bevacizumab, Capecitabine and Cisplatin vs Placebo, Capecitabine and Cisplatin; Test type: Superiority or Other; p = 0.4709, Log Rank; The difference in distribution of progression-free survival between the two treatment arms was tested with a two-sided unstratified log-rank test; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.66 to 1.21] — The hazard ratio between the two treatment arms was estimated with a univariate Cox's proportional hazards model

5. Secondary Outcome: Percentage of Participants With PFS Events (Disease Progression/Death) During First-line Therapy
Description: Progression of disease was defined as at least 20% increase in the sum of longest diameters of target lesions compared to the smallest sum of longest diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. PFS during first-line therapy was defined as the time between randomization and the date of first documented disease progression or death, whichever occurred first and only if it occurred no later than 28 days after last confirmed intake of any study medication and before the start of non-study antineoplastic treatment, according to RECIST.
Time Frame: From randomization until disease progression or death (up to 26 months)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
percentage of participants | 51.0 | 59.8

6. Secondary Outcome: PFS During First-line Therapy
Description: PFS during first-line therapy was defined as time between randomization and date of first documented disease progression or death, whichever occurred first and only if it occurred no later than 28 days after last intake of any study medication and only if it occurred before start of non-study antineoplastic treatment, according to RECIST. Progression of disease was defined as at least 20% increase in sum of longest diameters of target lesions compared to smallest sum of longest diameters on-study & absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. PFS was estimated using Kaplan Meier method. Reported data included censored observations. Participants who neither progressed nor died in this interval, or who were lost to follow-up were censored at date of last tumor assessment/last follow-up within this time window. Participants for whom no post-baseline tumor assessments were available were censored at day of randomization.
Time Frame: From randomization until disease progression or death (up to 26 months)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
months | 6.3 [5.7 to 7.5] | 6.1 [5.5 to 7.6]
Statistical Analysis 1: Comparison: Bevacizumab, Capecitabine and Cisplatin vs Placebo, Capecitabine and Cisplatin; Test type: Superiority or Other; p = 0.3685, Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.58 to 1.22] — The hazard ratio between the two treatment arms was estimated with a univariate Cox's proportional hazards model

7. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Progression of disease was defined as at least 20% increase in the sum of longest diameters of target lesions compared to the smallest sum of longest diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: From randomization until disease progression or death (up to 26 months)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
percentage of participants | 56.0 | 53.9

8. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time between randomization and the first occurrence of disease progression. Progression of disease was defined as at least 20% increase in the sum of longest diameters of target lesions compared to the smallest sum of longest diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. Time to progression was estimated using Kaplan Meier method. Reported data included censored observations. Participants who had not progressed at the time of study completion (including participants who had died before disease progression) or who were lost to follow-up were censored at the date of the last tumor assessment or last follow-up for progression of disease. Participants for whom no post-baseline tumor assessments were available were censored at day of randomization.
Time Frame: From randomization until disease progression or death (up to 26 months)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
months | 6.5 [5.7 to 7.5] | 7.0 [5.8 to 8.5]
Statistical Analysis 1: Comparison: Bevacizumab, Capecitabine and Cisplatin vs Placebo, Capecitabine and Cisplatin; Test type: Superiority or Other; p = 0.8589, Log Rank; The difference in distribution of disease progression between the two treatment arms was tested with a two-sided unstratified log-rank test; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.67 to 1.41] — The hazard ratio between the two treatment arms was estimated with a univariate Cox's proportional hazards model

9. Secondary Outcome: Percentage of Participants With Best Overall Response as Assessed by RECIST During First-Line Therapy
Description: Best overall response during first-line therapy was defined as the occurrence of either a confirmed complete (CR) or a partial response (PR), as assessed by the RECIST criteria. CR: disappearance of all target and non-target lesions (TLs) and normalization of tumor markers. Pathological lymph nodes must have short axis measures less than (<) 10 mm. PR: at least a 30 % decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of TLs, taking as reference the baseline sum of longest diameters.
Time Frame: From randomization until disease progression or death (up to 26 months)
Population: Measurable disease population included all randomized participants who had measurable disease at baseline according to RECIST.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 81 | 86
percentage of participants | 40.7 [29.9 to 52.2] | 33.7 [23.9 to 44.7]
Statistical Analysis 1: Comparison: Bevacizumab, Capecitabine and Cisplatin vs Placebo, Capecitabine and Cisplatin; Test type: Superiority or Other; p = 0.3480, Chi-squared; Difference in Response Rates = 7.02, 95% CI 2-sided [-8.3 to 22.4] — Approximate 95% CI for difference of two rates using Hauck-Anderson method

10. Secondary Outcome: Duration of Response During First-Line Therapy
Description: Duration of response during first-line therapy was defined as the time from when response (CR or PR) was first documented to first documented disease progression or death (whichever occurs first) during first-line therapy. CR: disappearance of all target and non-TLs and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. PR: at least a 30 % decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of TLs, taking as reference the baseline sum of longest diameters. Duration of response was estimated using Kaplan Meier method. Reported data included censored observations. Participants who did not progress or die after they had had a confirmed response were censored at the date of their last tumor measurement or last follow-up for progression of disease during first line therapy.
Time Frame: From randomization until disease progression or death (up to 26 months)
Population: Measurable disease population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 81 | 86
months | 7.2 [4.9 to 11.3] | 5.8 [4.6 to 6.6]
Statistical Analysis 1: Comparison: Bevacizumab, Capecitabine and Cisplatin vs Placebo, Capecitabine and Cisplatin; Test type: Superiority or Other; p = 0.0462, Log Rank; The difference in distribution of response between the two treatment arms was tested with a two-sided unstratified log-rank test; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.29 to 1.00] — The hazard ratio between the two treatment arms was estimated with a univariate Cox's proportional hazards model

11. Secondary Outcome: Percentage of Participants With Disease Control During First-Line Therapy
Description: Disease control was defined as stable disease(SD) for 6 weeks or longer, CR plus PR as assessed by RECIST criteria for participants with measurable disease.CR:disappearance of all TLs & normalization of tumor markers. Pathological lymph nodes must have short axis measures<10 mm. PR:at least 30% decrease in sum of measures(longest diameter for tumor lesions and short axis measure for nodes)of TLs, taking as reference baseline sum of longest diameters.SD:neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression taking as reference smallest sum of longest diameters on study. For participants without measurable disease, clinical benefit rate was defined as no clinical disease progression for >/=6 weeks. Disease progression was defined as at least 20% increase in sum of diameters of TLs compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: From randomization until disease progression or death (up to 26 months)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
percentage of participants | 73.0 [63.2 to 81.4] | 72.5 [62.8 to 80.9]
Statistical Analysis 1: Comparison: Bevacizumab, Capecitabine and Cisplatin vs Placebo, Capecitabine and Cisplatin; Test type: Superiority or Other; p = 0.9426, Chi-squared; Difference in Disease Control Rates = 0.45, 95% CI 2-sided [-12.4 to 13.3] — Approximate 95% CI for difference of two rates using Hauck-Anderson method

12. Secondary Outcome: Change From Cycle 1 in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 36 (QLQ-C30) Scale Over Time
Description: EORTC QLQ-C30 included global health status (GHS)/quality of life (QOL), functional scales (physical, role, cognitive, emotional, and social), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulties). Most questions used a 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used a 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores were averaged and transformed to 0-100 scale; a higher score for Global Qol/functional scales=better level of QoL/functioning, or a higher score for symptom scale=greater degree of symptoms.
Time Frame: From Cycle 1 until disease progression (up to 26 months)
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
scores on scale
  GHS/QOL | 1.24 [0.70 to 1.78] | 0.73 [0.15 to 1.31]
  Physical Funtioning | -0.89 [-1.66 to -0.12] | -0.99 [-1.77 to -0.21]
  Role Functioning | -0.65 [-1.46 to 0.17] | -0.37 [-1.19 to 0.46]
  Emotional Functioning | -0.22 [-0.87 to 0.44] | 0.19 [-0.47 to 0.85]
  Cognitive Functioning | -0.51 [-1.09 to 0.07] | -0.41 [-1.00 to 0.18]
  Social Functioning | -0.27 [-1.02 to 0.48] | 0.08 [-0.68 to 0.85]
  Fatigue | -0.36 [-1.14 to 0.43] | -0.27 [-1.07 to 0.53]
  Nausea and Vomiting | -0.82 [-1.26 to -0.38] | -0.55 [-1.05 to -0.05]
  Pain | -0.55 [-1.13 to 0.03] | -0.22 [-0.83 to 0.38]
  Dyspnoea | -0.10 [-0.48 to 0.27] | -0.07 [-0.47 to 0.32]
  Insomnia | -0.57 [-1.04 to -0.09] | 0.26 [-0.28 to 0.80]
  Appetite Loss | -0.65 [-1.25 to -0.05] | -1.17 [-1.83 to -0.51]
  Constipation | -0.14 [-0.62 to 0.34] | -0.02 [-0.58 to 0.54]
  Diarrhoea | -0.29 [-0.69 to 0.11] | 0.00 [-0.44 to 0.45]
  Financial Difficulties | 0.31 [-0.57 to 1.19] | 0.04 [-0.86 to 0.94]

13. Secondary Outcome: Change From Cycle 1 in EORTC QLQ-STO22 Scale Over Time
Description: The EORTC QLQ-STO22 is a gastric cancer quality of life questionnaire. There are 22 questions which comprise 5 scales (dysphagia, pain, reflux symptom, dietary restrictions, and anxiety) and 4 single items (dry mouth, hair loss, taste, body image). Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 1 question was a yes or no answer). A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100; higher score=better level of functioning or greater degree of symptoms.
Time Frame: From Cycle 1 until disease progression (up to 26 months)
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Number analyzed (Participants) | 100 | 102
scores on scale
  Dysphagia | -0.31 [-0.63 to 0.02] | -0.05 [-0.40 to 0.30]
  Pain | -0.97 [-1.50 to -0.43] | -0.52 [-1.07 to 0.03]
  Reflux Symptoms | -0.27 [-0.78 to 0.24] | -0.43 [-0.95 to 0.09]
  Eating Restrictions | -0.30 [-0.75 to 0.15] | -0.36 [-0.83 to 0.10]
  Anxiety | -0.17 [-0.91 to 0.57] | -0.73 [-1.48 to 0.03]
  Dry Mouth | -0.19 [-0.94 to 0.55] | 0.68 [-0.08 to 1.44]
  Taste | -0.44 [-1.05 to 0.16] | -0.66 [-1.29 to -0.02]
  Body Image | 0.27 [-0.52 to 1.05] | 0.13 [-0.68 to 0.94]
  Hair Loss | -0.35 [-1.29 to 0.58] | -0.61 [-1.73 to 0.50]

ADVERSE EVENTS:
Time Frame: From randomization up to 26 months
Description: Safety population included all randomized participants who received at least one dose/infusion of any component of study medication.
Arm/Group | Bevacizumab, Capecitabine and Cisplatin | Placebo, Capecitabine and Cisplatin
Serious Adverse Events (participants affected / at risk) | 19/100 | 21/101
Other Adverse Events (participants affected / at risk) | 94/100 | 95/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, Capecitabine and Cisplatin (N=100) | Placebo, Capecitabine and Cisplatin (N=101)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 7
Intestinal obstruction (Gastrointestinal disorders) | 4 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastropleural fistula (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Lung infection (Infections and infestations) | 3 | 0
Fungal infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Death (General disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, Capecitabine and Cisplatin (N=100) | Placebo, Capecitabine and Cisplatin (N=101)
Nausea (Gastrointestinal disorders) | 59 | 56
Vomiting (Gastrointestinal disorders) | 61 | 53
Constipation (Gastrointestinal disorders) | 18 | 24
Diarrhoea (Gastrointestinal disorders) | 14 | 12
Abdominal pain (Gastrointestinal disorders) | 14 | 9
Abdominal distension (Gastrointestinal disorders) | 7 | 9
Neutropenia (Blood and lymphatic system disorders) | 38 | 40
Leukopenia (Blood and lymphatic system disorders) | 31 | 35
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 14
Anaemia (Blood and lymphatic system disorders) | 6 | 13
Granulocytopenia (Blood and lymphatic system disorders) | 3 | 6
Neutrophil count decreased (Investigations) | 29 | 28
White blood cell count decreased (Investigations) | 15 | 24
Platelet count decreased (Investigations) | 19 | 13
Haemoglobin decreased (Investigations) | 10 | 10
Aspartate aminotransferase increased (Investigations) | 7 | 6
Alanine aminotransferase increased (Investigations) | 6 | 6
Blood bilirubin increased (Investigations) | 7 | 4
Creatinine renal clearance decreased (Investigations) | 1 | 6
Decreased appetite (Metabolism and nutrition disorders) | 32 | 36
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 4
Fatigue (General disorders) | 24 | 24
Pyrexia (General disorders) | 14 | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 17 | 9
Hypertension (Vascular disorders) | 12 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Headache (Nervous system disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.